CLINICAL TRIAL: NCT03313414
Title: Hepatitis C Virus Post-Exposure Prophylaxis for Health Care Workers
Brief Title: HCV Post-Exposure Prophylaxis for Health Care Workers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participant enrollment, funding withdrawn.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Raymond Chung, Director of Hepatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017P001661
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis C
Keywords: HCV; Needlestick
MeSH Terms: conditions — Hepatitis C; Needlestick Injuries | interventions — Sofosbuvir; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Sofosbuvir/Velpatasvir (Experimental): 14 days of treatment with Sofosbuvir/Velpatasvir tablet
  Interventions: Drug: Sofosbuvir/Velpatasvir Treatment for 14 days

INTERVENTIONS:
Drug: Sofosbuvir/Velpatasvir Treatment for 14 days — 14 day therapy with Sofosbuvir/Velpatasvir
  Other Names: Epclusa

SUMMARY:
This is an unblinded, observational trial of sofosbuvir-velpatasvir in adult health care workers who are exposed to hepatitis C virus from needlestick injury with hollow-bore needles.

DETAILED DESCRIPTION:
The goal of this study is to assess the safety and tolerability of the use of sofosbuvir-velpatasvir in the setting of post-exposure prophylaxis among Health Care Workers exposed to HCV from needlestick injury with hollow-bore needles

ELIGIBILITY:
Inclusion Criteria:

* Healthcare worker with exposure through needlestick injury with hollow-bore needles to source patients who are HCV positive
* Healthcare worker must be HCV Ab-

Exclusion Criteria:

* HCV Ab positive
* HCV Ab negative and HCV RNA greater than 1000 IU/ml
* Active malignancy
* Positive urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Undetectable HCV RNA | 12 weeks post treatment
  Negative HCV viral RNA at 12 weeks after the last dose of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
no plan currently to share IPD with other researchers